CLINICAL TRIAL: NCT03166852
Title: Compliance to HIT-program at Home With the Use of Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Anne-Mette Dissing, Senior lecturer, PhD-fellow, University College of Northern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FOU-PHD-005
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2; Exercise; Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: One group performs HIT with techology-based feedback for 5 weeks and the next group do the same
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-training group (Experimental): High-intensity training at home 3 times/week for 5 weeks
  Interventions: Other: Home-training

INTERVENTIONS:
Other: Home-training — 5 weeks of interval training at home. The training consisted of 3 minutes of warm-up. 10 intervals of 1 minute at 90% of maxHR interspersed with one minute of low intensity pedalling. Cool-down period of 2 minutes.

SUMMARY:
High-intensity training (HIT) has showed beneficial effects in type 2 diabetics such as improved glycemic control, improved bloodpressure and more. In addition, HIT is a time-saving training protocol which is of importance, as lack of time often is mentioned as a reason not to train. The combination of the time-saving HIT-protocol and the possibility to train at home and still get feedback on the intensity and amount of training can be appealing for some. This study aims to investigate whether it is possible to train at the right intensity and frequency and only get feedback throug a technology.

DETAILED DESCRIPTION:
Participants:

Patients with diagnosed type 2 diabetes recruited through local papers and Facebook. The participants receives both oral and written information before signing a written consent.

Pretest Each participant participate in a 1½ hour long pretest in which basic information is collected. This information include gender, age, weight, height, diabetes-age, marital status, medicine and education/job. Furthermore they complete two questionnaires; the Diabetes Attitude Scale(DAS) and Health Literacy. The pretest-session ends with a VO2max test to find the participants maximal heart rate and their maximal oxygen consumption. Before leaving an appointment is made on when to get a visit at home with the purpose to get instructions on how to train and get the equipment.

DAS The questionnaire consisted of 33 statements divided into subgroups. The participant is instructed to consider each statement in terms of how much they agree with the statement and they is instructed to answer all the questions. A higher score overall indicates a positive attitude towards diabetes and the result can also be viewed as results in subgroups.

Health Literacy Health Literacy is found using the Danish TOFHLA (Test Of Functional Health Literacy in Adults). The Danish TOFHLA consists of a 17-item numeracy part and 50-item reading comprehension part. The numeracy part of the Danish TOFHLA assesses the participant's ability to understand financial assistance, keep a clinical appointment, understand instructions for taking medication, etc. In the Danish TOFHLA, the test of reading comprehension is conducted as a modified cloze procedure in which random words are deleted from a reading passage (31). In this case, every fifth to seventh word is deleted in healthrelated reading passages, and the participant then selects the most fitting word from a list of four possible words. The total scores for the Danish TOFHLA test are divided into three levels: inadequate (score: 0-59), marginal (score: 60-74) and adequate (score 75-100).

VO2max Bicycle test to exhaustion with direct measurement of oxygen consumption by Breath-by-breath on Masterscreen CPX. Warm-up for 5 min. on 50-75 watt followed by incremental increase in intensity by 25 watt each minute until exhaustion. The test is qualified as a VO2max test if Respiratory Exchange Ratio (RER) exceeded 1,1. Otherwise it was categorized as a VO2peak.

Training The participants is instructed to train 3 times/week for 5 weeks. Before each training a HR-sensor (Polar H7 Smart Bluetooth) is applied and connected to Endomondo via their smartphone. The training consists of 10 x 60 sec work on a bike at an intensity of ~90% of max HR interspersed by 60 sec of recovery sessions. The HR used for training is calculated based on the max HR found by VO2max test at pretest.

Feedback At Mondays, Wednesdays and Fridays the participants gets feedback via Endomondo. The feedback focuses on the intensity and frequency of training. If no training is logged for a week the participant will be contacted through mail.

Interview At the end of the training period the equipment is obtained and a semi-structured interview performed and taped on a dictaphone (app). The interview is classified into three areas: The training, the use of the equipment and the feedback. The interview is then transcribed and analyzed in NVIVO.

A phenomenological approach is chosen as the interest is focused on the individuals experiences of the phenomenon and thereby describe the phenomenon

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 diabetics
* In possession of a smartphone Approval from own general practitioner

Exclusion Criteria:

* Conditions contraindicating high-intensity training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2016-11-27 (Actual); Study Completion 2016-11-27 (Actual)

PRIMARY OUTCOMES:
Intensity of training | Through study completion, an average of 5 weeks
  Is it possible for type 2 diabetics to reach a high intensity on their own?
Frequency of training | Through study completion, an average of 5 weeks
  How often do they train on their own?

SECONDARY OUTCOMES:
Diabetes Attitude Score | At baseline
  Questionaire to measure their attitude towards diabetes
Health Literacy | At baseline
  Questionaire
Interview | At study completion (After 5 weeks of training)
  A semi-structured interview evaluating experiences from the study, including the use of equipment, training-method etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ole K Hejlesen, Professor, Principal Investigator — Medical Informatics, Aalborg University, Denmark

IPD SHARING:
Plan to Share IPD: No